CLINICAL TRIAL: NCT01239303
Title: Effects of Citrulline on Gut Functioning During Excercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Kim van Wijck, MD, PhD student, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: MEC10-3-064
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Gastrointestinal; Hypoperfusion; Gut Damage
MeSH Terms: interventions — Citrulline; Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- citrulline (Active Comparator)
  Interventions: Dietary Supplement: Citrulline
- alanine (Placebo Comparator)
  Interventions: Dietary Supplement: alanine

INTERVENTIONS:
Dietary Supplement: Citrulline — single dose
  Arms: citrulline
Dietary Supplement: alanine — single dose
  Arms: alanine

SUMMARY:
During exercise, splanchnic perfusion is compromised, resulting in organ damage in healthy individuals. Improving the availability of NO might result increase splanchnic perfusion and prevent organ damage during exercise.

DETAILED DESCRIPTION:
The gastrointestinal (GI) tract plays an important role in the human body. The wall of the GI system regulates digestion and absorption of nutrients and it also has a very important function as a barrier between internal and external environment. The penetration of harmful substances and microbiota of the GI lumen (external environment) to the systemic circulation (internal environment) depends on this barrier. Previous studies have shown that exercise in healthy subjects provides hypoperfusion of the splanchnic area, resulting in intestinal damage, increased small intestinal permeability and liver damage. Similar splanchnic hypoperfusion occurs in patients with compromised circulation.

During episodes of splanchnic hypoperfusion, the de novo synthesis of nitric oxide (nitric oxide, NO) from arginine is compromised. This impaired NO synthesis may play a role in the development of organ dysfunction during exercise. L-citrulline administration, a precursor of arginine and NO, may result in improved NO availability and organ perfusion, thereby preventing organ damage.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18-35 years

Exclusion Criteria:

* not healthy
* use of medication or related products
* alcohol misuse
* smoking

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-01 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
GI perfusion | 2 hours
gut damage | 5 hours
microcirculation | 5 hours

SECONDARY OUTCOMES:
liver damage | 5 hours
kidney damage | 5 hours
amino acid analysis | 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands